CLINICAL TRIAL: NCT05216887
Title: A Randomized, Open-Label, Parallel-Arm Study to Assess the Pharmacokinetic Comparability of 2 Fixed Subcutaneous Doses of Aducanumab (BIIB037) With a Single, Weight-Based Intravenous Dose in Healthy Volunteers
Brief Title: A Study to Assess the Pharmacokinetic (PK) Comparability of 2 Fixed Subcutaneous (SC) Doses of Aducanumab (BIIB037) With a Single, Weight-Based Intravenous (IV) Dose in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221HV104
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — aducanumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aducanumab IV (Active Comparator): Participants will receive a single weight-based dose of aducanumab via IV infusion on Day 1.
  Interventions: Biological: Aducanumab
- Aducanumab SC (Experimental): Participants will receive 2 fixed doses of aducanumab via SC injection on Days 1 and 15.
  Interventions: Biological: Aducanumab

INTERVENTIONS:
Biological: Aducanumab — Administered as specified in the treatment arm.
  Other Names: BIIB037; Aduhelm

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetic (PK) comparability of 2 fixed subcutaneous (SC) doses of aducanumab with a single, weight-based intravenous (IV) dose of aducanumab in healthy volunteers. The secondary objectives of the study are to assess the safety and tolerability of aducanumab administered SC in healthy volunteers and to characterize additional PK parameters of 2 fixed SC doses of aducanumab and a single, weight-based IV dose of aducanumab.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index between 18 and 30 kilograms per meter square (kg/m^2), inclusive
* Japanese participant has both biological parents and all 4 grandparents of Japanese descent
* Have a negative polymerase chain reaction test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) on Day -1

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator
* History of severe allergic, anaphylactic or systemic hypersensitivity reactions, or of any allergic reactions that in the opinion of the Investigator are likely to be exacerbated by aducanumab, the excipients contained in the formulation, and if appropriate, any diagnostic agents to be administered during the study
* History of, or positive test result at Screening for, human immunodeficiency virus
* History of hepatitis C infection or positive test result at Screening for hepatitis C virus antibody
* Symptoms consistent with SARS-CoV-2 infection, per the judgment of the Investigator, within 14 days prior to Day -1, including but not limited to fever (temperature > 37.5 degrees Celsius [°C]), sore throat, new and persistent cough, shortness of breath, diarrhea, muscle aches, or loss of taste or smell
* Current enrollment in any other drug, biological, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 30 days prior to Day -1, or 5 half-lives, whichever is longer
* Any immunization or vaccination given within 10 days prior to administration of study treatment and for 10 days after administration of study treatment
* Mini mental state examination score of < 27 at Screening

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of Aducanumab | Predose and at multiple time points post-dose up to Day 99

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 99
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.
Number of Participants with Clinically Significant Abnormal Vital Sign Values | Up to Day 99
Number of Participants with Clinically Significant Abnormal 12-Lead Electrocardiogram (ECG) Values | Day 1 and Day 99
Number of Participants with Clinically Significant Abnormal Laboratory Values | Up to Day 99
Area Under the Concentration-Time Curve From Time 0 to Time of the Last Measurable Concentration (AUClast) of Aducanumab | Predose and at multiple time points post-dose up to Day 99
Area Under the Concentration-Time Curve From Time 0 to 4 Weeks (AUC0-4wk) of Aducanumab | Predose and at multiple time points post-dose up to Day 28
Maximum Observed Concentration (Cmax) of Aducanumab | Predose and at multiple time points post-dose up to Day 99
Time to Reach Maximum Observed Concentration (Tmax) for Aducanumab Administered SC | Predose and at multiple time points post-dose up to Day 99
Elimination Half-Life (t1/2) of Aducanumab | Predose and at multiple time points post-dose up to Day 99
Volume of Distribution (Vd) or Apparent Volume of Distribution (V/F) of Aducanumab | Predose and at multiple time points post-dose up to Day 99
Clearance (CL) or Apparent Clearance (CL/F) of Aducanumab | Predose and at multiple time points post-dose up to Day 99

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, Anaheim, California
  - QPS-MRA, Miami, Florida
  - QPS Missouri, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org